CLINICAL TRIAL: NCT03286842
Title: A Phase IIIb, Single-arm, Open-label Multicentre Study of Olaparib Monotherapy in the Treatment of HER2-ve Metastatic Breast Cancer Patients With Germline or Somatic BRCA1/2 Mutations.
Brief Title: To Study Clinical Effectiveness and Safety of Olaparib Monotherapy in Metastatic Breast Cancer Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00018
Record Dates: First submitted 2017-08-17; First posted 2017-09-19 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: HER2-ve Metastatic Breast Cancer; Germline BRCA1/2 Mutations; Somatic BRCA1/2 Mutations
Keywords: HER2-ve metastatic breast cancer; Germline BRCA1/2 mutations; Somatic BRCA1/2 mutations; BRCA1; BRCA2
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Olaparib 150mg tablets administered orally twice daily continuously
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Patients will be administered olaparib orally, twice daily at 300 mg. Two (2) 150 mg olaparib tablets should be taken at the same time each morning and evening of every day, approximately 12 hours apart.

SUMMARY:
This open-label, multi-centre phase IIIb study will assess the effectiveness, benefits and potential harms in the use of olaparib monotherapy treatment for patients with HER2-ve metastatic breast cancer associated with germline or somatic breast cancer susceptibility gene (gBRCA1/2 or sBRCA1/2) mutations.

DETAILED DESCRIPTION:
The study is a phase IIIb, multicenter, single-arm, open-label study designed to evaluate the clinical effectiveness in a real-world setting of olaparib monotherapy in patients with confirmed germline or somatic breast cancer susceptibility gene (gBRCA1/2 or sBRCA1/2) mutations. This study will generate additional data to support other olaparib studies, which may help inform and guide clinical practice. Physician defined the progression-free survival (PFS) for gBRCAm patients is the primary outcome measure. Based on the prevalence of gBRCA1/2 mutations, it is estimated that up to 1400 patients may require screening in order to identify 250 gBRCA mutated patients and 20 sBRCA mutated patients. Patients will be administered two olaparib 150mg tablets in morning and evening of every day after a light meal. Dose reductions may be required for olaparib treatment related toxicities. Patients should continue to receive study treatment until documented physician-defined disease progression as assessed by the investigator (gBRCA mutated patients), RECIST1.1 disease progression (sBRCA mutated patients) or unacceptable toxicity, or for as long as they do not meet any other discontinuation criteria. A positive benefit/risk profile is expected and no ethical issues are identified from exposing patients to olaparib within the planned clinical study.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent prior to any study specific procedures. For patients aged <20 years and screened in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative.
2. Patients must be ≥18 years of age.
3. Histologically or cytologically confirmed HER2-ve breast cancer with evidence of metastatic disease. Patients can have either TNBC (defined as oestrogen receptor and progesterone receptor negative [immunohistochemistry nuclear staining <1%] and HER2-ve [immunohistochemistry 0, 1+ or 2+ and/or in situ hybridization nonamplified with ratio less than 2.0]) or oestrogen receptor / progesterone receptor positive breast cancer as long as they are HER2-ve.
4. Documented BRCA1/2 status

   * To be regarded as BRCA1/2 (+ve), the patient must have a mutation that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental / lead to loss of function). Mutations that are not clearly pathogenic may be assessed by a committee of genetic specialists to adjudicate if the patient is eligible.
   * Patients with tBRCA mutations: must be confirmed by a validated method (e.g. results from a CLIA-certified laboratory or CE-IVD device)
5. Prior treatment with a taxane or an anthracycline in either an adjuvant (may include neoadjuvant) or metastatic breast cancer treatment setting.
6. Patients should have received no more than two prior cytotoxic chemotherapy regimens in the metastatic setting. If a patient has oestrogen receptor and/or progesterone receptor positive HER2 negative metastatic breast cancer and has completed a prior line of hormonal treatment, then if the current or currently planned choice of treatment for the patient does not include a hormonal treatment then they would be a suitable patient to enter the study. Previous endocrine therapy could be in either an adjuvant or a metastatic setting and include endocrine therapy in combination with a targeted agent such as a CDK4/6 or mTOR inhibitor.
7. Be considered suitable, by the Investigator, for further treatment with single-agent chemotherapy for the metastatic disease
8. Patients must have normal organ and bone marrow function measured within 14 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless the patient has documented Gilbert's Syndrome
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) / alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase (SGPT)) ≤ 2.5 x institutional ULN unless liver metastases are present in which case they must be ≤ 5x ULN
   * Patients must have creatinine clearance (CrCl) estimated using the Cockcroft- Gault equation of ≥ 51 mL/min or 24 hour urine test may be done if standard of care:

   Estimated CrCl = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72

   a- where F=0.85 for females and F=1 for males
9. Patients must have a life expectancy ≥ 16 weeks
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1

    Postmenopausal is defined as (at least one criterion met):
    * amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
    * luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range for women under 50
    * radiation-induced oophorectomy with last menses >1 year ago
    * chemotherapy-induced menopause with >1 year interval since last menses
    * surgical sterilisation (bilateral oophorectomy or hysterectomy).
11. Women of childbearing potential, who are sexually active, must agree to the use of one highly effective form of contraception and their male partners must use a condom from the signing of the informed consent, throughout the period of taking study treatment and for at least 1 month after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse.
12. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use one highly effective form of contraception if they are of childbearing potential.
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations for greater than 6 months.

Exclusion criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Exposure to an investigational product (IP) during the last 1 month or 5 half-lives (whichever is longer) prior to enrolment
4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
5. Any previous treatment with a PARP inhibitor, including olaparib
6. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
7. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
8. Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
9. Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
10. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
11. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML
12. Patients with symptomatic uncontrolled brain metastases.

    - Exception: Patients with adequately treated brain metastases documented by baseline CT or MRI scan that has not progressed since previous scans and that does not require corticosteroids (except ≤10 mg/day prednisone or equivalent for at least 14 continuous days prior to dosing) for management of CNS symptoms are eligible, provided that a repeat CT or MRI following the identification of CNS metastases (obtained at least 2 weeks after definitive therapy) must document adequately treated brain metastases.
13. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.

    Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
15. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
16. Breastfeeding women
17. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
18. Patients with a known hypersensitivity to olaparib or any of the excipients of the product
19. Patients with known active hepatitis (i.e., hepatitis B or C)
20. Whole blood transfusions in the last 28 days prior to entry to the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gelmon, MD, FRCPC, Principal Investigator — BritishColumbiaCancerAgency, 600W.10th Ave,Vancouver,Canada.
Locations (107):
- United States (2):
  - Research Site, Towson, Maryland
  - Research Site, Jackson, Mississippi
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- France (21):
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Quentin
  - Research Site, Toulouse
- Germany (8):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Hanover
  - Research Site, München
  - Research Site, Münster
  - Research Site, Rostock
- Research Site, Budapest, Hungary
- Italy (12):
  - Research Site, Aviano
  - Research Site, Bologna
  - Research Site, Candiolo
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Prato
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (3):
  - Research Site, Nagoya
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
- Poland (8):
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Grzepnica
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (9):
  - Research Site, Irkutsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Surgut
  - Research Site, Ufa
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam
  - Research Site, Seoul
- Spain (12):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Pamplona
  - Research Site, San Cristóbal de La Laguna
  - Research Site, Seville
  - Research Site, Vigo
  - Research Site, Zaragoza
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Mersin
  - Research Site, Tekirdağ
- United Kingdom (8):
  - Research Site, Cardiff
  - Research Site, Colchester
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Balmana J, Fasching PA, Couch FJ, Delaloge S, Labidi-Galy I, O'Shaughnessy J, Park YH, Eisen AF, You B, Bourgeois H, Goncalves A, Kemp Z, Swampillai A, Jankowski T, Sohn JH, Poddubskaya E, Mukhametshina G, Aksoy S, Timcheva CV, Park-Simon TW, Anton-Torres A, John E, Baria K, Gibson I, Gelmon KA; LUCY investigators. Clinical effectiveness and safety of olaparib in BRCA-mutated, HER2-negative metastatic breast cancer in a real-world setting: final analysis of LUCY. Breast Cancer Res Treat. 2024 Apr;204(2):237-248. doi: 10.1007/s10549-023-07165-x. Epub 2023 Dec 19. PMID 38112922
- [Derived] Gelmon KA, Fasching PA, Couch FJ, Balmana J, Delaloge S, Labidi-Galy I, Bennett J, McCutcheon S, Walker G, O'Shaughnessy J; Collaborating Investigators. Clinical effectiveness of olaparib monotherapy in germline BRCA-mutated, HER2-negative metastatic breast cancer in a real-world setting: phase IIIb LUCY interim analysis. Eur J Cancer. 2021 Jul;152:68-77. doi: 10.1016/j.ejca.2021.03.029. Epub 2021 Jun 1. PMID 34087573
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00018&attachmentIdentifier=aef63c74-06df-40d3-abe9-b750920e9fa5&fileName=D0816C00018_CSP_30Nov2020_Redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00018&attachmentIdentifier=c5f3b35e-e777-40b3-9b87-c363966f11d8&fileName=D0816C00018_SAP_30Nov2020_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00018&attachmentIdentifier=bf42d8ab-9b06-40de-a996-38cd1a8317d8&fileName=D0816C00018_Redacted_CSRSynopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 17-January-2018 to 21-March-2019 in 125 sites in 15 countries.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment. A total of 256 participants were enrolled in this study but, only 255 started treatment.
Groups:
- Olaparib: Participants received olaparib 300 mg tablets per dose level orally twice daily continuously given as 2 x 150 mg twice daily.
Period: Overall Study
Arm/Group | Olaparib
Started | 255
Completed | 175
Not Completed | 80
Not completed — Patients rolled over to another study | 80

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set consisted of all participants who received at least one dose of study treatment.
Arm/Group | Olaparib
Number analyzed (Participants) | 255
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed in both the rows sums up to the overall number.
  years
    Germline BRCA1/2 mutation (gBRCAm) cohort: number analyzed (Participants) | 252
    Germline BRCA1/2 mutation (gBRCAm) cohort | 46.2 (11.30)
    Somatic BRCA1/2 mutation (sBRCAm) cohort: number analyzed (Participants) | 3
    Somatic BRCA1/2 mutation (sBRCAm) cohort | 55.3 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in both the rows sums up to the overall number.
  Participants
    gBRCAm cohort: number analyzed (Participants) | 252
    gBRCAm cohort: Female | 248
    gBRCAm cohort: Male | 4
    sBRCAm cohort: number analyzed (Participants) | 3
    sBRCAm cohort: Female | 3
    sBRCAm cohort: Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in both the rows sums up to the overall number.
  Participants
    gBRCAm cohort: number analyzed (Participants) | 252
    gBRCAm cohort: Hispanic or Latino | 13
    gBRCAm cohort: Not Hispanic or Latino | 189
    gBRCAm cohort: Unknown or Not Reported | 50
    sBRCAm cohort: number analyzed (Participants) | 3
    sBRCAm cohort: Hispanic or Latino | 0
    sBRCAm cohort: Not Hispanic or Latino | 1
    sBRCAm cohort: Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in both the rows sums up to the overall number.
  Participants
    gBRCAm cohort: number analyzed (Participants) | 252
    gBRCAm cohort: American Indian or Alaska Native | 1
    gBRCAm cohort: Asian | 22
    gBRCAm cohort: Native Hawaiian or Other Pacific Islander | 0
    gBRCAm cohort: Black or African American | 2
    gBRCAm cohort: White | 177
    gBRCAm cohort: More than one race | 0
    gBRCAm cohort: Unknown or Not Reported | 50
    sBRCAm cohort: number analyzed (Participants) | 3
    sBRCAm cohort: American Indian or Alaska Native | 0
    sBRCAm cohort: Asian | 1
    sBRCAm cohort: Native Hawaiian or Other Pacific Islander | 0
    sBRCAm cohort: Black or African American | 0
    sBRCAm cohort: White | 0
    sBRCAm cohort: More than one race | 0
    sBRCAm cohort: Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in Real-world Setting in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting through assessment of PFS in germline BRCA mutated patients was evaluated. PFS is defined as the time from first dose of olaparib to the date of progression or death from any cause. In this study, disease progression in gBRCAm patients will be based on Investigator assessment, i.e. radiological ( e.g. RECIST) progression, symptomatic progression, or clear progression of non-measurable disease, as long as progression can be documented.
Time Frame: At every visit until the earliest of disease progression, death or end of study (up to 3 years)
Population: The Full Analysis Set consisted of all participants who received at least one dose of study treatment. The number analyzed in both the rows sums up to the overall number.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Olaparib gBRCAm Cohort: Participants received olaparib 300 mg tablets orally twice daily continuously given as 2 x 150 mg twice daily.
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 8.18 [6.97 to 9.17]

2. Secondary Outcome: Overall Survival (OS) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of overall survival in germline BRCA mutated participants was determined. OS is defined as the time from first dose of olaparib to the date of death from any cause.
Time Frame: At every visit and until death or end of study (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 24.94 [21.06 to 28.91]

3. Secondary Outcome: Time to First Subsequent Treatment or Death (TFST) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of time to use of subsequent therapies, second progression, and study treatment discontinuation in germline BRCA mutated participants was determined. TFST is defined as the time from first dose of olaparib to first subsequent treatment commencement or death if this occurs before commencement of first subsequent treatment.
Time Frame: At every visit until start of first subsequent anticancer treatment or death or end of study (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 9.40 [8.61 to 10.64]

4. Secondary Outcome: Time to Second Subsequent Treatment or Death (TSST) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of time to use of subsequent therapies, second progression, and study treatment discontinuation in germline BRCA mutated participants was determined. TSST is defined as the time from first dose of olaparib to second subsequent treatment commencement or death if this occurs before commencement of second subsequent treatment.
Time Frame: At every visit until start of second subsequent anticancer treatment or death or end of study (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 14.72 [13.50 to 17.25]

5. Secondary Outcome: Time to Study Treatment Discontinuation or Death (TDT) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of time to use of subsequent therapies, second progression, and study treatment discontinuation in germline BRCA mutated patients was determined. TDT is defined as the time from first dose of olaparib to study treatment discontinuation or death if this occurs before discontinuation of study treatment.
Time Frame: At every visit and until discontinuation of study treatment or death or end of study (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 7.98 [6.90 to 8.54]

6. Secondary Outcome: Time to Second Progression or Death (PFS2) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of time to use of subsequent therapies, second progression, and study treatment discontinuation in germline BRCA mutated participants was determined. PFS2 is defined as the time from first dose of olaparib to the earliest progression event subsequent to that used for the primary variable PFS or death from any cause. Patients alive and for whom a second disease progression has not been observed will be censored at the last time known to be alive and without a second disease progression. In this study, disease progression in gBRCAm patients will be based on Investigator assessment, i.e. radiological ( e.g. RECIST) progression, symptomatic progression, or clear progression of non-measurable disease, as long as progression can be documented
Time Frame: At every visit until second progression or death or end of study (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
months | 14.49 [13.17 to 17.05]

7. Secondary Outcome: Clinical Response Rate (CRR) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of clinical response rate and duration of clinical response in germline BRCA mutated participants was determined. CRR is defined as the percentage of patients assessed by the Investigator as responding. Response in gBRCAm patients were based on the Investigator's assessment. Data obtained up until progression, or last evaluable assessment in the absence of progression, will be included in the assessment of CRR. However, any responses, which occurred after a further anticancer therapy was received, will not be included in the numerator for the CRR calculation.
Time Frame: At every visit until disease progression or death or end of study (up to 3 years)
Population: The Full Analysis Set consisted of all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
Percentage of participants | 49.6 [43.3 to 55.9]

8. Secondary Outcome: Duration of Clinical Response (DoCR) in Germline BRCA Mutated Participants
Description: The clinical effectiveness of olaparib treatment in HER2-ve metastatic breast cancer participants in a real-world setting by assessment of clinical response rate and duration of clinical response in germline BRCA mutated participants was determined. DoCR is defined as the time from the date the Investigator first assessed the patient as responding to the date the Investigator assessed the patient as progressing or the date of death from any cause. The end of response should coincide with the date of progression or death used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing towards the first visit response. If a patient does not progress following a response, they will be censored at the PFS censoring date.
Time Frame: At every visit until disease progression or death or end of study (up to 3 years)
Population: The Full Analysis Set consisted of all participants who received at least one dose of study treatment.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Olaparib gBRCAm Cohort
Number analyzed (Participants) | 252
Months | 8.0 [4.2 to 18.6]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The safety and tolerability of olaparib treatment in HER2-ve metastatic breast cancer patients in a real-word setting was evaluated.
Time Frame: From Screening (Day -28 to Day -1) until post DCO [up to 3 years]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Olaparib sBRCAm Cohort: Participants received olaparib 300 mg tablets per dose level orally twice daily continuously given as 2 x 150 mg twice daily.
Arm/Group | Olaparib gBRCAm Cohort | Olaparib sBRCAm Cohort
Number analyzed (Participants) | 252 | 3
Participants
  Any AE | 243 | 3
  Any AE casually related to study treatment | 214 | 3
  Any AE of CTCAE grade 3 or higher | 69 | 2
  Any AE of CTCAE grade 3 or higher, causally related to study treatment | 44 | 1
  Any AE with outcome = death | 0 | 0
  Any AE with outcome = death, causally related to study treatment | 0 | 0
  Any SAE (including events with outcome = death) | 32 | 1
  Any SAE (including events with outcome = death), causally related to study treatment | 10 | 0
  Any AE leading to discontinuation of study treatment | 16 | 0
  Any AE leading to discontinuation of study treatment, causally related to study treatment | 11 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -28 to -1) until post DCO [up to 3 years].
Arm/Group | Olaparib gBRCAm Cohort | Olaparib sBRCAm Cohort
All-Cause Mortality (participants affected / at risk) | 140/252 | 2/3
Serious Adverse Events (participants affected / at risk) | 32/252 | 1/3
Other Adverse Events (participants affected / at risk) | 243/252 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib gBRCAm Cohort (N=252) | Olaparib sBRCAm Cohort (N=3)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (4) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (10) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib gBRCAm Cohort (N=252) | Olaparib sBRCAm Cohort (N=3)
Nasopharyngitis (Infections and infestations) | 14 (17) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (22) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 98 (168) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 22 (37) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 41 (71) | 1 (6)
Decreased appetite (Metabolism and nutrition disorders) | 31 (36) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (15) | 0 (0)
Dizziness (Nervous system disorders) | 23 (28) | 0 (0)
Dysgeusia (Nervous system disorders) | 16 (18) | 0 (0)
Headache (Nervous system disorders) | 47 (103) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (40) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 21 (25) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 19 (31) | 0 (0)
Constipation (Gastrointestinal disorders) | 30 (37) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 53 (72) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 25 (30) | 0 (0)
Nausea (Gastrointestinal disorders) | 140 (236) | 2 (2)
Vomiting (Gastrointestinal disorders) | 67 (111) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (55) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (32) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (24) | 0 (0)
Asthenia (General disorders) | 70 (94) | 2 (3)
Fatigue (General disorders) | 59 (84) | 0 (0)
Pyrexia (General disorders) | 31 (43) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03286842/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT03286842/SAP_001.pdf